CLINICAL TRIAL: NCT06588621
Title: HEalthCAre Workers' Health: a Transversal Evaluation
Acronym: HECATE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240415; 2024-A00383-44 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Occupational Health
Keywords: Occupational health; Mental health; Occupational medicine; Resident
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Residents at Cochin Port Royal Hospital: Residents at Cochin Port Royal Hospital assessed by the occupational health department during the analysis period (November 2023- October 2025).
  Interventions: Other: Questionnaire on physical and mental health among healthcare professionnals

INTERVENTIONS:
Other: Questionnaire on physical and mental health among healthcare professionnals — Feedback on the results of the questionnaire and toolkit on resources with regard to healthy habits in the professional setting

SUMMARY:
The research focuses on assessing the overall health of residents at the Cochin Port Royal hospital Group.

* physical health
* Mental health: detection of signs of anxiety, depression, eating disorders, substance abuse, etc.
* Sexual health
* Quality of medical care (dental, gynecological)
* Knowledge of risk prevention, particularly infectious risks, in the workplace.

DETAILED DESCRIPTION:
In the societal and medical crisis the investigators are currently facing, healthcare workers are a key element in maintaining public health institutions.

Nevertheless, their health has only been analyzed and managed from a fragmented or piecemeal perspective, despite the multiple dimensions of their health vulnerabilities: physical health, mental health, eating disorders, sedentary lifestyles, risk behaviours and so on.

In 2022, the occupational medicine department at Hôpital Cochin-Port-Royal will be systematically evaluating all residents during their 6-month internship at the hospital (not just new residents, during their first internship at AP-HP). To the knowledge of the investigators, this initiative is unique among AP-HP hospitals.

The investigators hope to take advantage of this unique procedure to gain a more precise knowledge of the health of residents at AP-HP in 2023-5.

The primary objective is to evaluate the health status of residents in a tertiary teaching hospital.

Secondary objectives:

* Determine the relevance and performance of a systematic occupational health consultation offered to every resident at the center.
* Identify levers for improvement to meet the unmet health needs of this specific population.

ELIGIBILITY:
Inclusion Criteria:

- Residents at Cochin Port Royal hospital between November 2023 and October 2025

Exclusion Criteria:

* Opposition to anonymous data collection
* Residents who benefited from the evaluation outside the analysis period: November 2023-October 2025.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents at Cochin Port Royal hospital between November 2023 and October 2025
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Residents | Up to 17 months
  Percentage of Residents presenting at least one of the following disorders: anxiety, depression, burnout, eating disorders, drug misuse, risk behaviours, reported drug use.

SECONDARY OUTCOMES:
Number of residents | Up to 17 months
  Number of residents assessed in occupational medicine / number of salaried residents.
Percentage of Residents | Up to 17 months
  Percentage of residents with no GP, no gynaecological check-up, no proven chronic pathology and not up to date with vaccinations.
Percentage of Residents | Up to 17 months
  Percentage of each disorder among residents: anxiety syndrome, depression, burnout, eating disorders, drug misuse, risk behaviors, reported substance abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Charlier, MD, PhD, Study Director — Infectious diseases department of Cochin hospital
Locations (1):
- Cochin University Hospital, Paris, IDF, France

REFERENCES:
- [Background] Bai X, Wan Z, Tang J, Zhang D, Shen K, Wu X, Qiao L, Zhou Y, Wang Y, Cheng W, Jiang W, Wang L, Tian X. The prevalence of burnout among pulmonologists or respiratory therapists pre- and post-COVID-19: a systematic review and meta-analysis. Ann Med. 2023 Dec;55(1):2234392. doi: 10.1080/07853890.2023.2234392. PMID 37459584
- [Background] Metse AP, Clinton-McHarg T, Skinner E, Yogaraj Y, Colyvas K, Bowman J. Associations between Suboptimal Sleep and Smoking, Poor Nutrition, Harmful Alcohol Consumption and Inadequate Physical Activity ('SNAP Risks'): A Comparison of People with and without a Mental Health Condition in an Australian Community Survey. Int J Environ Res Public Health. 2021 Jun 1;18(11):5946. doi: 10.3390/ijerph18115946. PMID 34206135
- [Background] Ghotbi N, Pilz LK, Winnebeck EC, Vetter C, Zerbini G, Lenssen D, Frighetto G, Salamanca M, Costa R, Montagnese S, Roenneberg T. The microMCTQ: An Ultra-Short Version of the Munich ChronoType Questionnaire. J Biol Rhythms. 2020 Feb;35(1):98-110. doi: 10.1177/0748730419886986. Epub 2019 Dec 3. PMID 31791166
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychol Med. 1982 Nov;12(4):871-8. doi: 10.1017/s0033291700049163. PMID 6961471
- [Background] Chaltiel D, Adjibade M, Deschamps V, Touvier M, Hercberg S, Julia C, Kesse-Guyot E. Programme National Nutrition Sante - guidelines score 2 (PNNS-GS2): development and validation of a diet quality score reflecting the 2017 French dietary guidelines. Br J Nutr. 2019 Aug 14;122(3):331-342. doi: 10.1017/S0007114519001181. Epub 2019 Jul 25. PMID 31342885
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Ewing JA. Detecting alcoholism. The CAGE questionnaire. JAMA. 1984 Oct 12;252(14):1905-7. doi: 10.1001/jama.252.14.1905. PMID 6471323
- See also: Related Info — http://beh.santepubliquefrance.fr/beh/2019/13/2019_13_1.html
- See also: Related Info — https://drees.solidarites-sante.gouv.fr/publications/rapports/enquete-nationale-perinatale-2016-les-naissances-et-les-etablissements
- See also: Related Info — https://www.has-sante.fr/upload/docs/application/pdf/2010-10/corriges_synthese_carie_dentaire_version_postcollege-10sept2010.pdf
- See also: Related Info — https://www.scirp.org/reference/referencespapers?referenceid=1146501